CLINICAL TRIAL: NCT04504474
Title: Network Analysis of Co-morbid Symptoms of Adult Major Depressive Disorder and Attention-deficit Hyperactivity Disorder in an Outpatient Population
Brief Title: Network Analysis of Adult MDD and ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Health Sciences North Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 18-056
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is an investigation to determine co-morbid symptoms between adult major depressive disorder (MDD) and adult attention-deficit hyperactivity disorder (ADHD) using a novel statistical technique called network analysis.

ELIGIBILITY:
Inclusion Criteria:

* participants have a diagnosis of MDD or ADHD or both
* participants are competent to consent to the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will gather a recruitment of 500 male and female outpatients from the Psychiatric Outpatient Clinic at Kirkwood Site attached to Health Sciences North.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-08-08 (Estimated); Study Completion 2021-09-08 (Estimated)

PRIMARY OUTCOMES:
Co-morbidity | September 8, 2021
  Characterize the ADHD/MDD symptom network in a psychiatric outpatient setting comprised of adults
Network reliability | September 8, 2021
  Determine the stability and reliability of this network
Central symptoms | September 8, 2021
  Determine the central symptoms that lead to co-activation of ADHD/MDD clusters

CONTACTS AND LOCATIONS:
Locations (1):
- Kirkwood Site - Health Sciences North, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
None of the IPD will be shared with other researchers